CLINICAL TRIAL: NCT02309645
Title: A Prospective Randomized Controlled Study Evaluating the Safety and Efficacy of EVICEL® Used for Suture-Line Sealing in Dura-Mater Closure During Paediatric Neurosurgical Cranial Procedures
Brief Title: The Paediatric EVICEL® Neuro Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study completed the required elements (40 paediatric subjects) per regulatory requirement. The study enrolled 40/42 subjects. No safety signals were identified. No changes required to the statistical analysis as described in the protocol.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOS-13-006; 2013-003558-26 (EudraCT Number)
Record Dates: First submitted 2014-10-02; First posted 2014-12-05 (Estimated); Results first posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2022-08

CONDITIONS: CSF Leak
Keywords: fibrin sealant; CSF leak
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVICEL® Fibrin Sealant (Experimental): EVICEL® is a human plasma-derived fibrin sealant. EVICEL® consists of two components: a concentrate of Human Clottable Protein (referred to as Biological Component 2; BAC2) and a solution of Human Thrombin. No material of animal origin is present in the product
  Interventions: Biological: EVICEL® Fibrin Sealant
- Sutures Only (Other): Subjects randomized to control will receive additional dural repair sutures as deemed necessary by the surgeon to attempt to achieve a watertight closure.
  Interventions: Other: Sutures Only

INTERVENTIONS:
Biological: EVICEL® Fibrin Sealant — Subjects randomized to receive EVICEL® Fibrin Sealant (Human), a thin layer will be applied to the entire length of the suture line and the adjacent area to at least 5mm away, including all suture holes.
  Other Names: EVICEL, fibrin sealant
  Arms: EVICEL® Fibrin Sealant
Other: Sutures Only — Subjects randomized to Control (Additional Sutures) will receive additional dural repair sutures applied immediately to the dural suture line after randomization as deemed necessary by the surgeon.
  Arms: Sutures Only

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of EVICEL® when used for suture-line sealing in dura-mater closure in elective or urgent paediatric cranial neurosurgery to provide intraoperative watertight closure.

DETAILED DESCRIPTION:
This is a prospective randomized, open-label, multi-center controlled study evaluating the effectiveness of EVICEL® as an adjunct to sutured dural closure compared to control to obtain an intraoperative watertight dural closure.

Paediatric subjects, undergoing elective or urgent craniotomy/craniectomy for pathological processes in the posterior fossa (such as benign or malignant tumors, vascular malformations, and Chiari 1 malformations) or in the supratentorial region and who were demonstrated to have persistent cerebrospinal fluid (CSF) leakage following a primary attempt at suture closure of the dural incision.

Paediatric subjects for this study are classified as:

* Newborn infants (birth to 27 days. Pre-term newborn infants born ≤ 37 weeks gestation will be included within the group)
* Infants and toddlers (28 days to <24 months)
* Children (2 to 11 years)
* Adolescents (12 to <18 years)

  42 paediatric subjects with intra-operative cerebrospinal fluid (CSF) leak following primary suturing of the dura will be randomized in a 2:1 allocation ratio and will be stratified by surgical procedure, posterior fossa or supratentorial to either EVICEL® Fibrin Sealant (Human) or additional dural sutures.

Subjects will be followed post-operatively through discharge and for 30 days (±3 days) post-surgery. The incidence of CSF leaks will be assessed within 5 days (± 2 days) and 30 days (±3 days) post-operatively as detected by any of the following: clinical observation, diagnostic testing or the need for surgical intervention to treat a CSF leak or pseudomeningocele.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective or urgent craniotomy/craniectomy for pathological processes in the posterior fossa (such as benign or malignant tumors, vascular malformation, and Chiari 1 malformations) or in the supratentorial region and who are demonstrated to have persistent CSF leakage following primary attempt at suture closure of the dural incision;
* Administration of perioperative antibiotic prophylaxis;
* Patients who are less than 18 years of age;
* Patients who are able and willing to comply with the procedures required by the protocol;
* The subject's parent/legal guardian must be willing to give permission for the subject to participate in the trial, and provide written informed consent for the subject. In addition, assent must be obtained from paediatric subjects who possess the intellectual and emotional ability to comprehend the concepts involved in the trial.
* Surgical wound classification Class I (refer to Appendix II). Penetration of mastoid air cells during partial mastoidectomy is permitted;
* The cuff of native dura along the craniotomy edge on each side is wide enough based on surgeon's judgment to facilitate suturing and to allow for sufficient surface area for adherence of the investigational product.

Exclusion Criteria:

* Subjects with a dura lesion from a recent surgery that still has the potential for CSF leakage;
* Conditions or treatments significantly compromising the immune system (such as AIDS);
* Known hypersensitivity to the components (human fibrinogen, arginine hydrochloride, glycine, sodium chloride, sodium citrate, calcium chloride, human thrombin, human albumin, mannitol and sodium acetate) of the investigational product;
* Hydrocephalus, except occlusive hydrocephalus caused by posterior fossa pathology to be treated.
* Existing CSF (ventricular, etc.) drains, shunts, Cushing/Dandy cannulation or Burr holes which damage the dura;
* Female subjects of childbearing potential with a positive urine or serum pregnancy test within 24 hours prior to surgery;
* Female subjects who are breastfeeding or intend to become pregnant during the clinical study period;
* Participation in another clinical trial with exposure to another investigational drug or device within 30 days prior to enrollment or expected during the study period;
* Scheduled or foreseeable surgery within the follow-up period.
* Dura injury during craniotomy/craniectomy that cannot be eliminated by widening the craniotomy/craniectomy to recreate the native dura cuff;
* Use of implants made of synthetic materials coming into direct contact with dura (e.g., PTFE patches, shunts, ventricular and subdural drains);
* Planned use of dural patches after primary suture closure of the dura;
* Placement of Gliadel Wafers;
* Persistent signs of increased brain turgor;
* Patient has a gap between durotomy edges of greater than 2mm after primary dural closure.
* Intersecting durotomy scars in the surgical path from a previous operation that cannot be completely removed by the planned dura resection;
* Two or more separate dura defects;
* Major intraoperative complications that require resuscitation or deviation from the planned surgical procedure.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (7):
- United Kingdom (7):
  - Clinical Investigation Site #24, Edinburgh
  - Clinical Investigation Site #22, Leeds
  - Clinical Investigation Site #21, Liverpool
  - St George's University Hospitals NHS Foundation Trust, London
  - Clinical Investigation Site #25, London
  - Clinical Investigation Site #23, Manchester
  - Clinical Investigation Site #20, Oxford

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sivakumar G, Magdum S, Aquilina K, Kandasamy J, Josan V, Ilie B, Barnett E, Kocharian R, Pettorini B. Safety and effectiveness of Evicel(R) fibrin sealant as an adjunct to sutured dural repair in children undergoing cranial neurosurgery. Childs Nerv Syst. 2024 Sep;40(9):2735-2745. doi: 10.1007/s00381-024-06434-4. Epub 2024 May 10. PMID 38727726

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was randomized to 'Sutures Only' arm but received EVICEL, and hence this participant was analyzed in the 'Sutures Only' arm for efficacy analysis (full analysis set [FAS]) and in the EVICEL arm for safety analysis.
Groups:
- EVICEL Fibrin Sealant: Participants who underwent craniectomy or craniotomy and had an intra-operative cerebrospinal fluid (CSF) leak, received up to 2 applications (maximum 4 layers) of EVICEL; applied to cover the entire length of the suture line and the adjacent area to at least 5 millimeters (mm) away, including all suture holes.
- Sutures Only (Control): Participants who underwent craniectomy or craniotomy and had an intra-operative CSF leak, received additional dural repair sutures as deemed necessary by the surgeon.
Period: Overall Study
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control)
Started | 26 | 14
Full Analysis Set (FAS) | 25 | 15
Completed | 26 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control) | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.4) | 9.2 (4.3) | 9.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 14 | 9 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success (Intraoperative Watertight Closure) in the Treatment of Intraoperative Cerebrospinal Fluid (CSF) Leakage
Description: Percentage of participants with success (intraoperative watertight closure) in the treatment of intraoperative CSF leakage were reported. Success is defined as no CSF leakage from dural repair intraoperatively, during Valsalva Maneuver 20-25 centimeters (cm) water (H2O) for 5-10 seconds.
Time Frame: Intraoperative (up to 1 day)
Population: The full analysis set (FAS) consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control)
Number analyzed (Participants) | 25 | 15
Percentage of participants | 92.0 | 33.3

2. Secondary Outcome: Number of Participants Experiencing CSF Leakage Within 7 Days Post-operatively
Description: Number of participants experiencing CSF leakage within 7 days post-operatively were reported.
Time Frame: Up to 7 days post-operatively
Population: The safety analysis set consisted of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control)
Number analyzed (Participants) | 26 | 14
Participants | 0 | 1

3. Secondary Outcome: Number of Participants Experiencing CSF Leakage Within 33 Days Post-operatively
Description: Number of participants experiencing CSF leakage within 33 days post-operatively were reported.
Time Frame: Up to 33 days post-operatively
Population: The safety analysis set consisted of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control)
Number analyzed (Participants) | 26 | 14
Participants | 0 | 1

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE (also referred to as an adverse experience) could be any unfavorable and unintended sign, symptom, or disease temporarily associated with the use of a drug, without judgment about causality. Since post-operative pain was an expected outcome of this type of surgery, for purposes of this study, only exacerbations of expected post-operative pain based on the investigator's judgment was reported as an AE.
Time Frame: Up to 33 days
Population: The safety analysis set consisted of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control)
Number analyzed (Participants) | 26 | 14
Participants | 22 | 14

5. Secondary Outcome: Number of Participants With Surgical Site Infections (SSI) According to National Healthcare Safety Network (NHSN) Criteria Within 33 Days Post-operatively
Description: Number of participants with SSI according to NHSN criteria within 33 days post-operatively were reported. NHSN CRITERIA states that infections occur within 33 days after the operation and infection involves only skin or subcutaneous tissue of the incision and at least one of the following: a) Purulent drainage, with or without laboratory confirmation, from the superficial incision; b) Organisms isolated from an aseptically obtained culture or fluid or tissue from the superficial incision; c) At least one of the following signs or symptoms of infection: pain or tenderness, localized swelling, redness, or heat and superficial incision is deliberately open by surgeon, unless incision is culture-negative; d) Diagnosis of superficial incisional SSI by the surgeon or attending physician.
Time Frame: Up to 33 days
Population: The safety analysis set consisted of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control)
Number analyzed (Participants) | 26 | 14
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 33 days
Description: The safety analysis set consisted of all participants who received treatment.
Arm/Group | EVICEL Fibrin Sealant | Sutures Only (Control)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/14
Serious Adverse Events (participants affected / at risk) | 5/26 | 8/14
Other Adverse Events (participants affected / at risk) | 22/26 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVICEL Fibrin Sealant (N=26) | Sutures Only (Control) (N=14)
Neurofibromatosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhagic cyst (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medulloblastoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 2 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Pneumocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVICEL Fibrin Sealant (N=26) | Sutures Only (Control) (N=14)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (2)
Dilatation ventricular (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Eye Swelling (Eye disorders) | 4 (4) | 4 (4)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 12 (14) | 6 (9)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 5 (8)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Implant site effusion (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 6 (6) | 3 (4)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 2 (2)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (11) | 5 (6)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Pneumocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT02309645/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02309645/SAP_001.pdf